CLINICAL TRIAL: NCT04692753
Title: Effect of Intensive Training and Education of Health Care Workers on the Maintenance of Venous Access Devices in Critically Ill Patients at a Tertiary Care Academic Hospital
Brief Title: Effect of Education of Health Care Workers on the Maintenance of Venous Access Devices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rubina Sharma, Junior Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: NK/6491/MD/147
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Vascular Access Devices
Keywords: intensive care unit; health care workers; central venous catheters
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-intervention: baseline data prior to training and education of health care workers. Intervention: intensive training and education of workers for maintenance of venous access devices.
- Post intervention: observation after training and education of health care workers
  Interventions: Other: Training and education

INTERVENTIONS:
Other: Training and education — Training and education of health care workers in the form of online seminars and bed side demonstration of care and maintenance of venous access devices
  Groups: Post intervention

SUMMARY:
In intensive care units (ICU), critically ill patients require various venous access devices for fluid resuscitation, drug therapy, or renal replacement therapy (RRT). These include peripheral intravenous catheters (PIVC), specialized venous ports like central venous catheters (CVCs), and hemodialysis ports. The investigators plan to do this pre- and post-intervention study to know the effect of intensive training and education of HCW (doctors and nurses) on the condition of venous access devices in critically ill patients.

DETAILED DESCRIPTION:
Phase 1, pre-intervention: The first twelve weeks will include 25 random visits to main ICU and point observations of all venous access devices under parameters like condition of dressing, connectors and documentation. This will also include the comparison of incidence of CLABSI in the pre and post intervention phase.

Phase 2, intervention: Next four weeks will be an intervention in the form of intensive training and education of the HCW (doctors and nurses). The intensive training will be in the form of an online presentation in which the investigators would have videos on care and maintenance of venous access devices, and the importance of documentation of days of insertion and change of dressing.

Phase 3, post-intervention: Another twelve weeks, post-intervention, again 25 random visits will be done to collect point observations about the same parameters of venous access devices and documentation as done in phase 1.

Statistical analysis: Each of these point observation parameters (for central or peripheral venous access) will be finally categorized as appropriate/inappropriate as per guidelines for best practice.

The compiled data from pre and post intervention phases would be compared. All the categorical parameters (appropriate/inappropriate) will be compared using chi-square test. All the quantitative parameters (e.g. incidence of CLABSI) will be compared using a paired t-test

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Main ICU

Exclusion Criteria:

* Patients who refuse to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to Main ICU of PGIMER during the period of data collection
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
To study the effect of intensive training and education of health care workers on care and maintenance of venous access devices in critically ill patients | Seven months
  the maintenance of venous access devices as evident from multiple point observations regarding condition of site ,dressing, connectors

SECONDARY OUTCOMES:
effect of intensive training and education on incidence of CLABSI during pre and post intervention phase | seven months
  incidence of central line associated blood stream infection to be compared between pre and post intervention phase

OTHER OUTCOMES:
to study improvement in documentation regarding venous access devices | seven months
  effect of training and education will be studied on improvement in documentation of venous access devices in post intervention phase

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No